CLINICAL TRIAL: NCT02210325
Title: An Open-Label, Randomized, Multi-Center Study to Evaluate the Efficacy and Safety of a Single Dose of Oral Solithromycin Compared to Single-Dose Intramuscular Ceftriaxone Plus Single-Dose Oral Azithromycin in the Treatment of Male and Female Patients With Uncomplicated Urogenital Gonorrhea With or Without Concomitant Chlamydia
Brief Title: Efficacy and Safety Study of Oral Solithromycin Compared to Intramuscular Ceftriaxone Plus Oral Azithromycin in the Treatment of Patients With Gonorrhea
Acronym: SOLITAIRE-U
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE01-302; 15-0091, HHSN272201300013 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Uncomplicated Urogenital Gonorrhea
Keywords: gonorrhea; chlamydia; solithromycin
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections | interventions — solithromycin; Ceftriaxone; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftriaxone plus Azithromycin (Active Comparator): A single intramuscular dose of 500 mg ceftriaxone plus a single oral dose of 1000 mg azithromycin
  Interventions: Drug: ceftriaxone; Drug: azithromycin
- Solithromycin (Experimental): A single oral dose of 1000 mg solithromycin
  Interventions: Drug: solithromycin

INTERVENTIONS:
Drug: solithromycin
  Arms: Solithromycin
Drug: ceftriaxone
  Arms: Ceftriaxone plus Azithromycin
Drug: azithromycin
  Arms: Ceftriaxone plus Azithromycin

SUMMARY:
This study will compare a single dose of oral solithromycin to the standard of care (intramuscular ceftriaxone plus oral azithromycin) in the treatment of patients with urogenital gonorrhea. A completed open-label Phase 2 study with single doses of solithromycin resulted in 100% microbiological eradication in male and female patients with uncomplicated urogenital gonorrhea.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 of the following:

  1. Untreated male with urethral gonorrhea as determined by a screening laboratory test (either NAAT or culture) for N. gonorrhoeae within 2 weeks prior to study drug administration.
  2. Untreated female with cervical gonorrhea as determined by a screening laboratory test (either NAAT or culture) for N. gonorrhoeae within 2 weeks prior to study drug administration.
  3. Urethral (male) or cervical (female) Gram stain demonstrating Gram-negative intracellular diplococci and leukocytes.
* The patient must be willing to abstain from anal, oral, and vaginal sexual intercourse or use condoms for all of these until study completion.
* Females of childbearing potential (including females less than 2 years post-menopausal) must have a negative pregnancy test at enrollment.

Exclusion Criteria:

* Confirmed or suspected complicated or systemic gonococcal infections such as pelvic inflammatory disease, epididymitis, arthritis, endocarditis, or disseminated gonococcal infection.
* Individuals who have already received antibiotic treatment for their gonorrhea.
* Use of systemic or intravaginal antibiotics within 7 days prior to study drug administration.
* Women who are pregnant or nursing.
* Men with suspected or confirmed rectal gonorrhea and symptoms of proctitis.
* History of significant intolerance or allergy to macrolide or cephalosporin antibiotics.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
To assess the eradication rate of Neisseria gonorrhoeae by culture following a single dose of oral solithromycin compared to single-dose intramuscular ceftriaxone plus oral azithromycin in the Microbiological Intent to Treat population. | 7 days after treatment

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single oral dose of solithromycin compared to single-dose IM ceftriaxone plus single-dose oral azithromycin in patients with gonorrhea | 7 days
  Adverse event frequency and severity will be compared between patients who received solithromycin and those who received ceftriaxone plus azithromycin
To compare bacterial eradication rates of N. gonorrhoeae from rectal or pharyngeal cultures following a single dose of oral solithromycin compared to single-dose IM ceftriaxone plus oral azithromycin. | 7 days
To assess clearance or persistence of N. gonorrhoeae and Chlamydia trachomatis nucleic acid from male and female genital, pharyngeal and rectal specimens. | 21 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Chen, MD, PhD, Principal Investigator — Melbourne Sexual Health Centre
Locations (5):
- United States (3):
  - Baltimore, Maryland
  - Cleveland, Ohio
  - Toledo, Ohio
- Australia (2):
  - Sydney, New South Wales
  - Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MY, McNulty A, Avery A, Whiley D, Tabrizi SN, Hardy D, Das AF, Nenninger A, Fairley CK, Hocking JS, Bradshaw CS, Donovan B, Howden BP, Oldach D; Solitaire-U Team. Solithromycin versus ceftriaxone plus azithromycin for the treatment of uncomplicated genital gonorrhoea (SOLITAIRE-U): a randomised phase 3 non-inferiority trial. Lancet Infect Dis. 2019 Aug;19(8):833-842. doi: 10.1016/S1473-3099(19)30116-1. Epub 2019 Jun 10. PMID 31196813